CLINICAL TRIAL: NCT03561038
Title: Randomized Trial Comparing the Franseen and Fork-top Needles for EUS-guided Fine-needle Biopsy of Solid Mass Lesions.
Brief Title: Comparing the Franseen and Fork-top Needles for EUS-guided Fine-needle Biopsy of Solid Mass Lesions.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar study just got done
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 217910
Record Dates: First submitted 2018-06-06; First posted 2018-06-19 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2019-04

CONDITIONS: Solid Mass Lesions in GI Tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Franseen Needle (Active Comparator): 2 strokes within the mass with Franseen Needle, and then 2 strokes with the Fork-tip Needle
  Interventions: Device: Franseen Needle
- Fork-tip Needle (Active Comparator): 2 strokes within the mass with Fork-Tip needle, and then 2 strokes with the Franseen Needle
  Interventions: Device: Fork-tip Needle

INTERVENTIONS:
Device: Franseen Needle — Comparing 2 needles designed for tissue acquisition
  Arms: Franseen Needle
Device: Fork-tip Needle — Comparing 2 needles designed for tissue acquisition
  Arms: Fork-tip Needle

SUMMARY:
This will be a randomized controlled trial of all the patients referred to University of Arkansas Medical for Medical Sciences (UAMS) for endoscopic ultrasound (EUS) guided biopsy of solid mass lesions. EUS guided tissue acquisition will be performed in all these patients using both needle types (22-gauge Franseen Fine Needle Biopsy (FNB) (Acquire, Boston Scientific Corporation, Natick, Mass) and 22-gauge Fork-tip FNB needle (SharkCore, Medtronic)) with randomization of the order in which the needle will be used.

DETAILED DESCRIPTION:
All procedures will be performed by the advance endoscopists Dr Sumant Inamdar (SI) and Dr Benjamin Tharian (BT) using a linear array echoendoscope (Olympus UCT180, Olympus America Corp, Center Valley, Pa) with patients in the left lateral decubitus position after administration of anesthesia (propofol or general anesthesia). During EUS, the mass will first be punctured using either needle based on the randomization assignment. Tissue acquisition will be performed using the fanning maneuver (4 strokes at 4 different locations within the mass). After performing 2 dedicated passes for cell block for histological analysis using the randomized needle, 2 additional passes will be made for cell block with the alternate needle. Sample obtained from each pass is placed into a separate container to be analysed separately. The occurrence of immediate adverse events will be noted at the time of procedure, and late adverse events will be documented by follow-up telephone calls at 1 week post-procedure

ELIGIBILITY:
Inclusion Criteria:

* Subjects from any ethnic background
* Successfully completes the screening process
* Has signed written informed consent by patient or surrogate
* Demonstrate willingness to follow protocol requirements, including follow-up schedule, and completion of study questionnaires.
* Patients must have evidence of a lesion seen on endoscopic ultrasound that is accessible
* Lack of severe or terminal co-morbidity, as judged by the generalists or specialists caring for the patient.

Exclusion Criteria:

* History of allergic reaction of hypersensitivity to the medications / anesthesia.
* Female participants of childbearing age who are pregnant
* Female participants who are breastfeeding.
* Participant has history of significant cardiovascular or pulmonary disease (e.g., myocardial infarct, unstable angina, congestive heart failure, arrhythmia, pulmonary edema or COPD), or other significant cerebrovascular disease (stroke)
* Patients who are uncooperative, unable to give written informed consent, who cannot return for follow-up, or refuse informed consent
* Persistent shock or hypertension (e.g., systolic blood pressure less than or equal to 99 mm mercury) that is unresponsive to less than or equal to 6 units of packed red blood cell (RBC) transfusions or requires continuous intravenous infusions of vasoactive drugs for blood pressure elevation.
* Severe coagulopathy unresponsive to blood transfusions (e.g., international normalized ratio >2.0, platelet count <20,000. activated partial thromboplastin time greater than 2.0 x normal, or bleeding time > 10 minutes)
* Contraindication to urgent endoscopy or follow-up procedures or inaccessible due to altered anatomy, moderate / tense ascites.
* Participant has uncontrolled diabetes / uncontrolled hypertension / severe immunodeficiency.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield | Up to 2 years
  comparing rates of diagnostic yield between the 2 cohorts.

SECONDARY OUTCOMES:
Histology | up to 2 years
  Histology will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Sumant Inamdar, MD, Principal Investigator — University of Arkansas

IPD SHARING:
Plan to Share IPD: No